CLINICAL TRIAL: NCT00183170
Title: Residual Effects of Intoxication on Student Performance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H-23064; P60AA013759 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Alcoholic Intoxication; Neurobehavioral Manifestations
Keywords: Alcohol abuse; Alcoholic beverages (beer); Residual effects; Psychomotor performance; Psychomotor vigilance test; Neurobehavioral Evaluation System; Family history of alcohol use; Alcoholic Consumption; Unhealthy alcohol use; Alcohol
MeSH Terms: conditions — Alcoholic Intoxication; Neurobehavioral Manifestations; Alcoholism | interventions — Ethanol; Beer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alcohol then Placebo (Experimental): Participants report for their first dosing night where they receive several alcohol drinks. After a wash out period of 1 week they then return and receive several placebo drinks. Participants sleep at the study site, are monitored overnight, and the next morning are awakened and escorted to the performance trials.
  Interventions: Drug: Alcohol; Other: Placebo
- Placebo then Alcohol (Experimental): Participants report for their first night where they receive several placebo drinks. After a wash out period of 1 week they then return and receive several alcohol drinks. Participants sleep at the study site, are monitored overnight, and the next morning are awakened and escorted to the performance trials.
  Interventions: Drug: Alcohol; Other: Placebo

INTERVENTIONS:
Drug: Alcohol — Participants report for their first dosing night where they receive several alcohol/beer drinks sufficient to raise their BrAC to 0.10 g%. Participants are breath-tested after completing their required dose. Participants return in a week for the 2nd session and receive placebo drinks. Participants are breath-tested after completing their placebo drinks.
  Other Names: Beer
Other: Placebo — Participants report for their first night where they receive several placebo drinks. Participants are breath-tested after completing their placebo drinks. Participants return in a week for the 2nd session and receive alcohol drinks sufficient to raise their BrAC to 0.10 g%. Participants are breath-tested after completing their required dose.
  Other Names: Non-alcoholic drink

SUMMARY:
The primary goal of the study is to assess the residual effects of heavy drinking on academic performance. The investigators will also explore whether these effects differ by family history of alcohol abuse and hangover symptoms, as well as compare males and females with respect to these effects. The primary hypothesis is that intoxication (0.10 g% blood alcohol concentration [BAC]) with an alcoholic beverage impairs next-day academic performance, as measured by scores on quizzes, standardized academic achievement tests, and standardized neurobehavioral assessments. The secondary hypothesis is that family-history-positive individuals will show a greater performance decrement the day after heavy drinking than family-history-negative individuals.

DETAILED DESCRIPTION:
The primary goal of the study is to assess the effect of heavy drinking on next day academic performance. A placebo-controlled 2-period crossover design will be used to compare the effects of dosing status on academic performance, with participants serving as their own controls. Participants are dosed on two separate occasions, once with non-alcoholic beverage and the other time with alcoholic beverage sufficient to raise blood alcohol to 0.10 g%. The morning after dosing, participants' academic performance is measured using a standardized achievement test (Graduate Record Exam). Participants' cognition is tested using the the Psychomotor Vigilance Test (PVT). Data on participants' demographics, family history of drinking problems and alcohol use. We are also collecting information on hangover symptoms and sleep quality the morning after dosing, in addition to participants' self ratings of academic performance. The procedure is conducted twice with one week in between, switching the individuals' dosing status, presenting a different, but comparable lecture and reading, and administering a different quiz based on the new lecture and reading and a different, but comparable standardized achievement exam. This design is intended to test the hypothesis that intoxication (0.10 g% BAC) with alcoholic beverage impairs next-day academic performance.

Participation involves a total of five sessions over a two week period. Participants are undergraduates who volunteer and meet inclusion criteria. Prior to enrollment, volunteers are screened to ensure they meet initial eligibility criteria. Eligible volunteers receive written instructions regarding participation and are scheduled for the study sessions. Participants report to the study site on the first session for an additional screening by the study physician and go through the informed consent process. Eligible participants report back the next week for their first dosing night where they receive several drinks (alcohol or placebo) sufficient to raise their Breath Alcohol Level (BrAC) to 0.10 g%; the amount of beverage administered is based on their body weight. Those receiving placebo receive the same total quantity of beverage as those receiving alcohol. Both alcohol-dosed and placebo-dosed participants are breath-tested after they have completed their required dose. Participants sleep at the study site and are monitored overnight. The next morning they are awakened and are escorted to the exam room for the performance trials. They return the next week for the second dosing night/dosing morning, and receive either alcohol or placebo, depending on what was administered the previous week, and take different but comparable performance tests.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-30
* Currently enrolled in college/university
* Have had 5 or more drinks (4 if female) in the last 30 days
* Score less than a 5 on the Short Michigan Alcohol Screening Test (SMAST)
* No self-reported history of counseling or treatment for substance abuse
* Not taking any medication contraindicated for alcohol use or that disrupts sleep
* Doesn't have a health condition contraindicated for alcohol use
* Has not been diagnosed with a primary sleep disorder
* Has not been diagnosed with a mental health disorder
* Not currently working night shifts at a job
* Not routinely taking medications that affect sleep
* If female, is using reliable birth control when necessary
* Not a regular smoker
* Likes the taste of beer

Exclusion Criteria:

* Less than age 21 and greater than age 30
* Not currently enrolled in college/university
* Hasn't had 5 or more drinks (4 if female) in the last 30 days (not a regular drinker)
* Score greater than or equal to 5 on the Short Michigan Alcohol Screening Test (SMAST)
* Self-reported history of counseling or treatment for substance abuse
* Taking any medication contraindicated for alcohol use or that disrupts sleep
* Has a health condition contraindicated for alcohol use
* Has been diagnosed with a primary sleep disorder
* Has been diagnosed with a mental health disorder
* Currently working night shifts at a job
* Routinely taking medications that affect sleep
* Is a regular smoker
* Is currently pregnant or nursing
* If female, is not using reliable birth control when necessary
* Not a regular drinker
* Dislikes the taste of beer

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howland, PhD MPH MPA, Principal Investigator — Boston University
Locations (1):
- General Clinical Research Center/Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohsenow DJ, Howland J, Winter M, Bliss CA, Littlefield CA, Heeren TC, Calise TV. Hangover sensitivity after controlled alcohol administration as predictor of post-college drinking. J Abnorm Psychol. 2012 Feb;121(1):270-5. doi: 10.1037/a0024706. Epub 2011 Aug 22. PMID 21859168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 239 participants were enrolled but 27 dropped out prior to randomization into the study arms so a total of 212 were randomized.
Period: First Intervention
Arm/Group | Alcohol, Then Placebo | Placebo, Then Alcohol
Started | 103 | 109
Completed | 101 | 109
Not Completed | 2 | 0
Not completed — Did not complete study | 1 | 0
Not completed — Did not meet targeted BrAC | 1 | 0
Period: Washout 1 Week
Arm/Group | Alcohol, Then Placebo | Placebo, Then Alcohol
Started | 101 | 109
Completed | 95 | 101
Not Completed | 6 | 8
Not completed — Did not complete study | 6 | 8
Period: Second Intervention
Arm/Group | Alcohol, Then Placebo | Placebo, Then Alcohol
Started | 95 | 101
Completed | 94 | 99
Not Completed | 1 | 2
Not completed — Did not complete study | 1 | 0
Not completed — Did not meet targeted BrAC | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol, Then Placebo | Placebo, Then Alcohol | Total
Number analyzed (Participants) | 94 | 99 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.46 (0.62) | 21.48 (0.66) | 21.47 (0.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 86
  Male | 49 | 58 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 80 | 155
  Black | 3 | 5 | 8
  Asian | 7 | 6 | 13
  Other | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 94 | 99 | 193
Maximum breath alcohol concentration (BrAC) [Mean (Standard Deviation); unit: g%] | 0.12 (0.01) | 0.12 (0.01) | 0.12 (0.01)
Amount of alcohol received [Mean (Standard Deviation); unit: ml] — Population: The mean and standard deviations of alcohol received for males and females differed so the results are stratified by sex.
  ml
    Males: number analyzed (Participants) | 49 | 58 | 107
    Males | 1607 (310) | 1611 (272) | 1609 (288)
    Females: number analyzed (Participants) | 45 | 41 | 86
    Females | 1137 (172) | 1106 (187) | 1122 (178)
Family history of alcohol problems [Count of Participants; unit: Participants]
  Yes | 28 | 43 | 71
  No | 64 | 55 | 119
  Adopted | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Residual Effects of Heavy Drinking
Description: This outcome will be measured by the afternoon total mood disturbance score. This is part of the Profile of Mood States Questionnaire (POMS). POMS is a 35 item instrument with Likert responses from 0 to 4 where 0=not at all and 4=extremely. Range of scores can be 0 to 140, lower scores are more favorable.
Time Frame: next day
Population: 153 POMS questionnaires were analyzed since 40 of the 193 participants did not return the POMS questionnaire by the next day.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Alcohol; Placebo: Results by beverage condition.
Arm/Group | Alcohol | Placebo
Number analyzed (Participants) | 153 | 153
scores on a scale | 4.3 (10.19) | 1.93 (8.39)

2. Secondary Outcome: Cognitive Function in Response to Heavy Drinking
Description: This outcome measure will be assessed using the Visual Span Test- Backwards (VST-B). This is the mean maximum span of words repeated backwards correctly. Higher scores are more favorable
Time Frame: next day
Population: Data were analyzed for 186 of the 193 participants since 7 did not complete the VST-B.
Measure: Mean (Standard Deviation); unit: backwards words
Arm/Group | Alcohol | Placebo
Number analyzed (Participants) | 186 | 186
backwards words | 5.41 (0.89) | 5.67 (1.16)

3. Secondary Outcome: Academic Function in Response to Heavy Drinking
Description: This outcome will be measured by the mean Graduate Record Exam (GRE) quantitative score. The quantitative score can range from 200-800. Higher scores are more favorable.
Time Frame: next day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol | Placebo
Number analyzed (Participants) | 193 | 193
score on a scale | 615.75 (98.92) | 612.38 (94.64)

4. Secondary Outcome: Reaction Time Affected by Residual Effects of Heavy Drinking
Description: This outcome will be measured with the Continuous Performance Test (CPT) for reaction time in mean milliseconds (ms). Lower reaction times are more favorable.
Time Frame: next day
Population: Data were analyzed for 187 of the 193 participants since 6 did not complete the CPT.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Alcohol | Placebo
Number analyzed (Participants) | 187 | 187
milliseconds | 378.77 (35.48) | 375.98 (35.82)

5. Secondary Outcome: Effectiveness of Psychomotor Vigilance Testing as a Fitness-for-duty Test
Description: This outcome will be assessed with the Psychomotor Vigilance Test (PVT) in median milliseconds. The 10-min PVT measures sustained or vigilant attention by recording response times to visual (or auditory) stimuli that occur at random inter-stimulus intervals. Lower number of milliseconds are associated with greater vigilant attention.
Time Frame: next day
Population: Data were analyzed for 190 of the 193 participants since 3 did not complete the PVT.
Measure: Median (Standard Deviation); unit: milliseconds of response time
Arm/Group | Alcohol | Placebo
Number analyzed (Participants) | 190 | 190
milliseconds of response time | 223.40 (22.81) | 218.57 (20.25)

ADVERSE EVENTS:
Arm/Group | Alcohol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/193 | 0/193
Other Adverse Events (participants affected / at risk) | 5/193 | 0/193
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcohol (N=193) | Placebo (N=193)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No